CLINICAL TRIAL: NCT06654414
Title: Project QUIT+: Adapting and Testing a Smoking Cessation Intervention for Transgender and Gender Expansive Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely by NIH action with the stated reason that the goals of the study no longer effectuate NIH priorities.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Director of Behavioral Medicine Program/Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-3; 1R21CA292185-01 (NIH)
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation; Depression; Anxiety; Nicotine Dependence; Gender Minority Stress
Keywords: Smoking Cessation; Smoking; Tobacco Use; Tobacco Use Disorder; Substance-Related Disorder; Nicotine; Anxiety; Depression; Transgender Individuals; Gender Expansive Individuals; Gender Minority Stress; Distress Tolerance; Quitting; Cognitive Behavioral Therapy
MeSH Terms: conditions — Smoking Cessation; Depression; Anxiety Disorders; Tobacco Use Disorder; Smoking; Tobacco Use; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRIDE QUIT (Experimental): Participants in this adapted intervention arm (n=30) will receive empirically-based, Cognitive-Behavioral therapy-based strategies, tailored for transgender and gender diverse (TGD) individuals, which aims to help participants quit smoking and address gender minority stressors, anxiety, depression, and improve distress tolerance.
  This intervention group will likely receive 6-10 active weekly sessions, with the quit day set around session 4-6. They will also receive transdermal nicotine patches (TNP) for a period of 8 weeks prior to the quit session.
  Interventions: Behavioral: PRIDE QUIT
- Enhanced Treatment As Usual (ETAU) (Active Comparator): Participants in this arm (n=30) will receive enhanced treatment as usual at Fenway Health. These participants will attend one session (brief counseling), will come to the clinic for weekly assessments only, and receive the option of transdermal nicotine patch (TNP) and referral to the Quit Line.
  Interventions: Behavioral: Enhanced Treatment As Usual (ETAU)

INTERVENTIONS:
Behavioral: PRIDE QUIT — This is an adapted behavioral intervention based on the integrated treatment for smoking cessation, anxiety, and depressed mood, known as QUIT, for persons with HIV. Through our treatment adaption process of QUIT (guided by Aim 1 and 2 data), PRIDE QUIT will be a Cognitive-Behavioral therapy-based intervention tailored for transgender and gender diverse (TGD) individuals, aimed at to helping participants quit smoking and address gender minority stressors, anxiety, depression, and improve distress tolerance.
  There will be three major assessments: baseline (T1), at the end of the intervention (T2), and a three-month follow-up visit (T3). This intervention group will likely receive 6-10 weekly sessions, with the quit day set around session 4-6. They will also receive transdermal nicotine patches (TNP) for a period of 8 weeks prior to the quit session.
  Arms: PRIDE QUIT
Behavioral: Enhanced Treatment As Usual (ETAU) — Brief counseling, the option of nicotine replacement therapy, and referral to the Quit Line.
  Arms: Enhanced Treatment As Usual (ETAU)

SUMMARY:
Smoking remains the leading preventable cause of death in the United States, and there are persistent and significant disparities in tobacco use among transgender and gender diverse (TGD) individuals. Stigma, discrimination, gender dysphoria, and other gender minority stressors likely contribute to these disparities, and the increased burden of gender minority stress may also be driving higher prevalence rates of anxiety and depression, both of which are more common among TGD individuals and among those who smoke relative to comparison samples. This study will (1) explore the ways in which gender minority stressors and associated anxiety and depression compromise smoking cessation among TGD individuals, identifying elements in an existing smoking cessation intervention that need to be adjusted to meet their unique needs; (2) adapt an existing smoking cessation intervention for TGD individuals; and (3) evaluate the feasibility and acceptability of the adapted intervention in a pilot randomized controlled trial.

DETAILED DESCRIPTION:
Despite the substantial decrease in the prevalence of smoking over the past 50 years, there are persistent and significant disparities in tobacco use among transgender and gender diverse (TGD) individuals. The prevalence of cigarette use in TGD individuals is 45.7 - 62.3%, compared to 39.8% in cisgender individuals. There are also disparities in e-cigarette use among TGD people relative to cisgender adults (26.5% vs. 5.5% in transgender and cisgender men, respectively). Transgender individuals may be particularly vulnerable to the consequences of tobacco use, as hormone therapy among those who smoke increases heart disease risk, and smoking may hinder recovery from gender-affirming surgeries. Stigma, discrimination, gender dysphoria, and other gender minority stressors contribute to tobacco use disparities. Enacted stigma and discrimination toward TGD individuals are common (reported by over 75% of participants in some samples), and experiencing stigma or discrimination increases the odds of current cigarette smoking, e-cigarette use/vaping, and dual use among TGD people. Gender dysphoria and gender minority stress may also lead to and/or exacerbate disparities in anxiety and depression, which are major impediments to smoking cessation that are more prevalent among TGD than cisgender individuals. Anxiety symptoms co- occur with smoking at high rates and significantly impair cessation success. Similarly, depressed mood and major depressive disorder, both more common among individuals who smoke than among those who do not, are associated with reduced odds of cessation. Therefore, gender minority stress and high prevalence rates of anxiety and depression render TGD individuals particularly vulnerable to smoking cessation difficulties. A tailored smoking cessation intervention that builds cognitive behavioral skills for cessation as well as reduces gender minority stress and associated anxiety and depression symptoms has strong potential to mitigate tobacco use disparities among TGD individuals. The investigators propose to adapt an existing smoking cessation intervention (known as QUIT) to address the unique needs of TGD people. In focus groups with TGD individuals who use tobacco (N = up to 32) and providers (N = 8), the investigators will explore the ways in which gender minority stressors and associated anxiety/depression compromise cessation as well as identify content in the current version of the QUIT intervention that does and does not meet their needs. Providers will also comment on anticipated implementation barriers. Following the ADAPT-ITT model, the qualitative data will inform the adaptation of the intervention. The investigators will then test the feasibility and acceptability of the adapted intervention (QUIT+) in a pilot RCT (N = 60); the investigators will also assess for signals of clinically meaningful change in biologically verified 7-day point prevalence abstinence, average number of cigarettes smoked, gender minority stress, anxiety and depression symptoms, and distress tolerance. If deemed to be feasible and acceptable, the intervention will be ready for a hybrid efficacy/effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* aged 18+
* self-reported difference between sex assigned at birth and gender identity
* current use of combustible cigarettes OR recent use of combustible cigarettes (defined as at least 5 cigarettes-per-day at some point within the past 6 months) OR current use of nicotine-containing e-cigarettes with use of combustible cigarettes in the past 6 months (defined as 5 cigarettes-per-day)
* English-speaking.

Exclusion Criteria:

* unable to provide informed consent
* current interfering untreated or unstable major health condition that is event during screening (e.g., active mania, current psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Acceptability | Through the end of treatment intervention, approximately 10 weeks
  Acceptability will be assessed via a questionnaire, completed after every other treatment session, that measures the 7 constructs of the acceptability of health care interventions framework: affective attitude, burden, ethicality, coherence, opportunity costs, perceived effectiveness, and self-efficacy. The intervention will be deemed acceptable if at least 75% of the participants rate 4+ items on the acceptability questionnaires with a 4 or a 5 on the Likert-style scale.
Feasibility | Through participants' enrollment, approximately 6 months
  Feasibility of the intervention is a primary outcome measure that will be calculated based on three assessments: (1) interventionist fidelity to the protocol (via a review of 10% of session recordings to determine whether key themes were addressed), (2) session attendance, and (3) participant retention at follow-up. Feasibility will be demonstrated if at least (1) 80% of the reviewed sessions address all key themes, (2) 75% of the participants attend at least half of all treatment sessions; and (3) 70% of the participants complete the 3-month follow-up.

SECONDARY OUTCOMES:
7-Day Point Prevalence Abstinence | At the end of treatment intervention (approx. 10 weeks post-baseline) and at 3-month follow-up (T3; approx. 6 months post-baseline)
  7-day point prevalence abstinence will be verified via expired-air carbon monoxide (CO) assessed with a Smokerlyzer, with 5ppm indicating abstinence (24 hours to two weeks). Because CO expired-air readings are significantly lower among users of e-cigarettes, abstinence for those using mostly e-cigarettes at baseline will be verified by cotinine assessment via a NicConfirm Mouth Swab Cotinine test (30 ng/ml indicates abstinence of 1-4 days).
Gender Minority Stress | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  Gender minority stress will be measured via the internal experience subscales of the Gender Minority Stress and Resilience Measure (GMSRM), including non-affirmation of gender identity, internalized transphobia, negative expectations, nondisclosure, community connectedness, and pride. Participants respond to each statement using a five-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree."
Average Number of Cigarettes Smoked Per Day In The Past Week | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  Average number of cigarettes smoked per day in the past week, assessed via the Time Line Follow-Back measure.
Nonbinary Distal Stress (Nbi-DMSS ) | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  The Nbi-DMSS was evaluated for validity and reliability in the current study and aimed to measure distal stressors experienced by nonbinary people. Participants were instructed "Please indicate whether you have experienced the following and if so, when the most recent occurrence was" with response options Never (1), Over a Year Ago (2), Within the past year, (3), Within the past six months (4),and NA (0) for the Discrimination and Harassment subscale items. Participants were instructed "Please indicate how frequently you have experienced the following in the past 6 months" with response options Never (1), Rarely (2), Occasionally (3), Often (4), Always/Daily (5), NA (0) for the remaining subscales. Higher and more frequent reported occurrence indicate worse outcomes.
Proximal Minority Stress (Nbi-PMSS) | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  The Nbi-PMSS was evaluated for validity and reliability in the current study and aimed to measure distal stressors experienced by nonbinary people. For the Internalized Invalidation, Internalized Nonbinary Negativity, and Internalized Burdensomeness subscales, participants were instructed "How much do you currently agree or disagree with the following statements?" Response options were on a 7-point Likert scale from Strongly disagree (1) to Strongly agree (7), with an NA option (0). For the remaining subscales participants were instructed "Please indicate how frequently you have experienced the following in the past 6 months" with response options Never (1), Rarely (2), Occasionally (3), Often (4), Always/Daily (5), NA (0). Higher and more frequent reported occurrence indicate worse outcomes.
Nonbinary Resilience (Nbi-RS) | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  The Nbi-RS aims to measure unique resilience factors experienced by nonbinary people. Participants are asked, "How much do you currently agree or disagree with the following statements?" Response options were on a 7-point Likert scale from Strongly disagree (1) to Strongly agree (7), with an NA option (0). All scales and subscales can be scored by taking the mean, with higher scores indicating better outcomes.
Severity of Nicotine Dependence | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  Severity of nicotine dependence will be assessed via the Fagerstrom Test for Cigarette Dependence. In scoring, items are summed to yield a total score of 0-10, with higher scores indicating a more intense physical dependence on nicotine.
Anxiety and Depressive Symptoms | At baseline assessment, end of treatment intervention (approx. 10 weeks post-baseline), and 3-month follow-up (T3; approx. 6 months post-baseline)
  Anxiety and depressive symptoms will be assessed by the Mood and Anxiety Symptom Questionnaire (MASQ). Likert style: 1 (not at all) to 5 (extremely); scores range from 24 to 120, with higher scores indicating greater levels of symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Conall M O'Cleirigh, PhD, Principal Investigator — Massachusetts General Hospital, Behavioral Medicine Program; Amelia Stanton, PhD, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - Massachusetts General Hopsital, Boston, Massachusetts
  - Boston University - Charles River Campus, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Based on the approved DSMP, we plan to only share deidentified data via a controlled access repository. No PHI, recordings, or unconsented human data will be made available to other investigators.
Supporting Information: Study Protocol, SAP
Time Frame: According to the approved DSMP, data will be uploaded at 6-monthly intervals.
Access Criteria: Any shared data will be stored in the NIH-approved controlled access repository, Cancer Data Service (CDS). Other qualified investigators, with authorized CDS access will have access to this data.